CLINICAL TRIAL: NCT02714764
Title: Evaluation of Outcome Metrics in Alexander Disease
Acronym: AxD Outcomes
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry); University of Wisconsin, Madison (Other); Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16-012649
Record Dates: First submitted 2016-02-19; First posted 2016-03-21 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Alexander Disease
Keywords: Alexander Disease
MeSH Terms: conditions — Alexander Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to define the natural history of Alexander Disease, a leukodystrophy that causes neurological dysfunction. Investigators will obtain clinical outcome assessments to measure how the disease affects a patient's gross motor, fine motor, speech and language function, swallowing, and quality of life. Specimens are collected to measure glial fibrillary acidic protein (GFAP) levels in cerebrospinal fluid (CSF) and blood. The data obtained from this study will be used for the design of future treatment trials.

DETAILED DESCRIPTION:
Participants will be asked to complete physical examinations including physical therapy, occupational therapy, speech and language therapy, neurocognitive and swallowing assessments. Patients (or caretakers) may be asked to complete questionnaires as well. Specimen collection is an optional procedure. The study asks for participants to return at least once yearly to repeat assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Alexander Disease

Exclusion Criteria:

* Other Leukodystrophies will not be enrolled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been diagnosed with Alexander Disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01-26 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in Gross Motor Function Over Time | Up to 10 years
  Total score and dimensional scores (rolling/supine, crawling/traveling, sitting, standing, and walking/running) will be calculated at each visit. Change in total and dimensional scores over time will be assessed.

SECONDARY OUTCOMES:
Change in the Bruininks-Oseretsky Test of Motor Proficiency Over Time | Up to 10 years
  Composite score and scores for the 4 sub-scales will be calculated at each visit. Change in composite and subscale scores over time will be assessed.

OTHER OUTCOMES:
Change in Peabody Developmental Motor Scales Over Time | Up to 10 years
  Composite score and 4 sub-scales (reflexes, stationary, locomotion, object manipulation) will be calculated at each visit. Change in composite and subscale scores over time will be assessed.
Change in Rosetti Infant-Toddler Language Scale Over Time | Up to 10 years
  Change in six sub-scales (Interaction-Attachment, Pragmatics, Gesture, Play, Language Comprehension, and Language Expression) will be assessed at each visit for age applicable patients.
Change in Swallowing Performance Over Time | Up to 10 years
  A clinical swallow evaluation will be performed and assessed for change annually using an ordinal classification scale based on performance.
Change in Clinical Evaluation of Language Fundamentals Over Time | Up to 10 years
  Changes in the comprehensive scores will be assessed at baseline and then annually at each visit which will be scheduled within ± 2 months around the specified time point, for up to 10 years
Change in Peabody Picture Vocabulary Test Over Time | Up to 10 years
  Changes in comprehensive scores will be assessed at baseline and then annually at each visit which will be scheduled within ± 2 months around the specified time point, for up to 10 years
Change in Goldman-Fristoe Test of Articulation Over Time | Up to 10 years
  Changes in standardized scores will be assessed at baseline and then annually at each visit which will be scheduled within ± 2 months around the specified time point, for up to 10 years
Change in Physical Health Quality of Life for Patients | Up to 10 years
  Surveys will be used as a composite measure to understand a patient's physical health and how it may change during their disease course. An aggregate measure of survey scores will be analyzed at baseline and end of study. Compass-31, PedsQL-Gastrointestinal Symptom Scales, Patient Global Impression of Change, Patient Global Impression of Severity, Alexander Disease Patient Domain Impression of Change, Alexander Disease Patient Domain Impression of Severity, Most Bothersome Symptom, PROMIS Pediatric Physical Function-Mobility-Short Form, PROMIS Pediatric Physical Function-Pain Interference-Short Form, PROMIS Pediatric Physical Function-Upper Extremity- Short Form, Pediatric Bowel Movement Scoring Tool-Child Supplement II (PBMST), Caregiver Priorities and Child Health Index of Life with Disabilities (CP Child), Emesis Frequency Ladder, Multiple Sclerosis Quality of Life (MSQoL-54)
Change in Physical Health Quality of Life for Parents/Caregivers | Up to 10 years
  Surveys will be used as a composite measure to understand a parents/caregiver physical health and how it may change during their child/spouse disease course. An aggregate measure of survey scores will be analyzed at baseline and end of study. Multiple Sclerosis Quality of Life (MSQoL-54)
Change in Mental Health Quality of Life for Patients | Up to 10 years
  Surveys will be used as a composite measure to understand a patient's mental health and how it may change during their disease course. An aggregate measure of survey scores will be analyzed at baseline and end of study. PedsQL Quality of Life Inventory, Multiple Sclerosis Quality of Life (MSQoL-54)
Change in Mental Health Quality of Life for Parents/Caregivers | Up to 10 years
  Surveys will be used as a composite measure to understand a parents/caregiver mental health and how it may change during their child/spouse disease course. An aggregate measure of survey scores will be analyzed at baseline and end of study. Multiple Sclerosis Quality of Life-54 (MSQoL-54), Hospital Anxiety and Depression Scale (HADS), and Euro-QoL 5 Dimensions (EQ5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Waldman, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and Samples will be shared with University of Wisconsin, Madison.
Supporting Information: ICF
Time Frame: Up to 10 years
Access Criteria: Dr. Albee Messing and Tracy Hagemann, PHD are listed in the HIPAA section of the approved informed consent.

REFERENCES:
- [Derived] Joung J, Gallison K, Sollee JJ, Vigilante N, Cooper H, Liu GW, Ballester L, Faig W, Waldman AT. Acquisition and Loss of Developmental Milestones and Time to Disease-Related Outcomes in Cerebral Alexander Disease. J Child Neurol. 2023 Dec;38(13-14):672-678. doi: 10.1177/08830738231210040. Epub 2023 Nov 3. PMID 37920915